CLINICAL TRIAL: NCT01376557
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of LX4211 in Combination With Metformin in Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: Safety and Efficacy of LX4211 With Metformin in Type 2 Diabetes Patients With Inadequate Glycemic Control on Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX4211.1-202-DM; LX4211.202 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A (Experimental)
  Interventions: Drug: 75 mg LX4211
- Treatment B (Experimental)
  Interventions: Drug: 200 mg LX4211
- Treatment C (Experimental)
  Interventions: Drug: 400 mg LX4211
- Treatment D (Experimental)
  Interventions: Drug: 200 mg LX4211
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 75 mg LX4211 — Subjects will receive 75 mg LX4211 once daily
  Arms: Treatment A
Drug: 200 mg LX4211 — Subjects will receive 200 mg LX4211 once daily.
  Arms: Treatment B
Drug: 400 mg LX4211 — Subjects will receive 400 mg LX4211 once daily.
  Arms: Treatment C
Drug: 200 mg LX4211 — Subjects will receive 200 mg LX4211 twice daily.
  Arms: Treatment D
Drug: Placebo — Subjects will receive placebo once daily.
  Arms: Placebo

SUMMARY:
This study is intended to assess the effect on HbA1c of different dose regimens of LX4211 in combination with metformin in subjects with Type 2 Diabetes Mellitus who have inadequate glycemic control on metformin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects between the ages of 18 to 75 years, inclusive
* Confirmed diagnosis of Type 2 diabetes mellitus
* Meet required laboratory values at screening, including fasting plasma glucose less than 270 mg/dL
* Stable dose of metformin monotherapy greater than 1500 mg/day for at least 8 weeks
* Willing and able to provide written informed consent
* Willing and able to maintain consistent dietary, physical activity, and sleeping patterns throughout the study

Exclusion Criteria:

* History of Type 1 diabetes mellitus, diabetic ketoacidosis, hyperosmolar nonketotic syndrome, or diabetes resulting from pancreatic disorder or secondary diabetes
* History of renal disease or clinically significant abnormal kidney function tests
* Presence of active hepatic disease or clinically significant abnormal liver function tests
* Subjects with a history of heart attack, severe/unstable angina, or coronary revascularization procedure within 6 months prior to study Day 1
* History of clinically significant cardiac arrhythmias within one year of study Day 1
* Subjects with congestive heart failure
* Subjects with uncontrolled Stage III hypertension
* Triglycerides >1000 mg/dL at Screening
* Known history of HIV or hepatitis C
* History of illicit drug or alcohol abuse with one year of study Day 1
* Have had 2 or more emergency room visits, doctor visits, or hospitalizations due to hypoglycemia within 6 months of study Day 1
* Use of any other investigational drug within 30 days of study Day 1
* Prior exposure to LX4211
* Use of any medication or herbal supplement for the purpose of weight loss
* Chronic use of any antidiabetic therapy other than metformin in the 3 months prior to study Day 1
* Use of corticosteroids within 2 weeks prior to study Day 1
* Major surgery within 6 months of study Day 1
* Subjects with any history of severe gastroparesis
* Inability or difficulty swallowing whole capsules or tablets
* Women who are pregnant or breast feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ikenna Ogbaa, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (51):
- United States (51):
  - Lexicon Investigational Site, Anaheim, California
  - Lexicon Investigational Site, Carmichael, California
  - Lexicon Investigational Site, Greenbrae, California
  - Lexicon Investigational Site, La Jolla, California
  - Lexicon Investigational Site, Northridge, California
  - Lexicon Investigational Site, Orange, California
  - Lexicon Investigational Site, Pismo Beach, California
  - Lexicon Investigational Site, Tarzana, California
  - Lexicon Investigational Site, Tustin, California
  - Lexicon Investigational Site, Denver, Colorado
  - Lexicon Investigational Site, Newark, Delaware
  - Lexicon Investigational Site, Edgewater, Florida
  - Lexicon Investigational Site, Miami, Florida
  - Lexicon Investigational Site, Orlando, Florida
  - Lexicon Investigational Site, West Palm Beach, Florida
  - Lexicon Investigational Site, Winter Park, Florida
  - Lexicon Investigational Site, Blue Ridge, Georgia
  - Lexicon Investigational Site, Savannah, Georgia
  - Lexicon Investigational Site, Lafayette, Indiana
  - Lexicon Investigational Site, Madisonville, Kentucky
  - Lexicon Investigational Site, Baton Rouge, Louisiana
  - Lexicon Investigational Site, Brockton, Massachusetts
  - Lexicon Investigational Site, Waltham, Massachusetts
  - Lexicon Investigational Site, Traverse City, Michigan
  - Lexicon Investigational Site, Olive Branch, Mississippi
  - Lexicon Investigational Site, Kansas City, Missouri
  - Lexicon Investigational Site, Omaha, Nebraska
  - Lexicon Investigational Site, Las Vegas, Nevada
  - Lexicon Investigational Site, Great Neck, New York
  - Lexicon Investigational Site, West Seneca, New York
  - Lexicon Investigational Site, Greensboro, North Carolina
  - Lexicon Investigational Site, Winston-Salem, North Carolina
  - Lexicon Investigational Site, Grand Forks, North Dakota
  - Lexicon Investigational Site, Canal Fulton, Ohio
  - Lexicon Investigational Site, Dayton, Ohio
  - Lexicon Investigational Site, Kettering, Ohio
  - Lexicon Investigational Site, Perrysburg, Ohio
  - Lexicon Investigational Site, Eugene, Oregon
  - Lexicon Investigational Site, Uniontown, Pennsylvania
  - Lexicon Investigational Site, Clinton, South Carolina
  - Lexicon Investigational Site, Mt. Pleasant, South Carolina
  - Lexicon Investigational Site, Chattanooga, Tennessee
  - Lexicon Investigational Site, Austin, Texas
  - Lexicon Investigational Site, Dallas, Texas
  - Lexicon Investigational Site, Houston, Texas
  - Lexicon Investigational Site, Killeen, Texas
  - Lexicon Investigational Site, San Antonio, Texas
  - Lexicon Investigational Site, Tomball, Texas
  - Lexicon Investigational Site, Ogden, Utah
  - Lexicon Investigational Site, Salt Lake City, Utah
  - Lexicon Investigational Site, Virginia Beach, Virginia

REFERENCES:
- [Derived] Rosenstock J, Cefalu WT, Lapuerta P, Zambrowicz B, Ogbaa I, Banks P, Sands A. Greater dose-ranging effects on A1C levels than on glucosuria with LX4211, a dual inhibitor of SGLT1 and SGLT2, in patients with type 2 diabetes on metformin monotherapy. Diabetes Care. 2015 Mar;38(3):431-8. doi: 10.2337/dc14-0890. Epub 2014 Sep 11. PMID 25216510

RESULTS

PARTICIPANT FLOW:
Groups:
- 75 mg LX4211 qd: Subjects will receive 75 mg LX4211 once daily
- 200 mg LX4211 qd: Subjects will receive 200 mg LX4211 once daily.
- 400 mg LX4211 qd: Subjects will receive 400 mg LX4211 once daily.
- 200 mg LX4211 Bid: Subjects will receive 200 mg LX4211 twice daily.
- Placebo qd: Placebo: Subjects will receive placebo once daily.
Period: Overall Study
Arm/Group | 75 mg LX4211 qd | 200 mg LX4211 qd | 400 mg LX4211 qd | 200 mg LX4211 Bid | Placebo qd
Started | 59 | 60 | 60 | 60 | 60
Completed | 51 | 54 | 55 | 54 | 53
Not Completed | 8 | 6 | 5 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 75 mg LX4211 qd | 200 mg LX4211 qd | 400 mg LX4211 qd | 200 mg LX4211 Bid | Placebo qd | Total
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 60 | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (9.61) | 55.6 (9.25) | 56.1 (9.51) | 56.4 (8.76) | 55.1 (9.79) | 55.9 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 43 | 31 | 31 | 34 | 164
  Male | 34 | 17 | 29 | 29 | 26 | 135
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 0 | 2
  Asian | 2 | 0 | 1 | 2 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 9 | 6 | 5 | 6 | 31
  White | 48 | 51 | 51 | 53 | 49 | 252
  More than one race | 1 | 0 | 1 | 0 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 14 | 21 | 12 | 15 | 82
  Not Hispanic or Latino | 39 | 46 | 39 | 48 | 45 | 217
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 59 | 60 | 60 | 60 | 60 | 299
Height [Mean (Standard Deviation); unit: cm] | 169.25 (10.419) | 166.99 (10.764) | 167.04 (9.849) | 169.39 (11.171) | 167.18 (10.240) | 167.96 (10.486)
Weight [Mean (Standard Deviation); unit: kg] | 96.16 (19.328) | 95.59 (19.368) | 91.38 (18.643) | 95.01 (22.202) | 90.57 (20.726) | 93.73 (20.093)
Body Mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.44 (5.237) | 34.23 (5.816) | 32.69 (5.757) | 32.85 (5.626) | 32.17 (5.796) | 33.08 (5.658)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c to Week 12
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | 75 mg LX4211 qd | 200 mg LX4211 qd | 400 mg LX4211 qd | 200 mg LX4211 Bid | Placebo qd
Number analyzed (Participants) | 56 | 58 | 57 | 57 | 57
% change | -0.42 (0.637) | -0.52 (0.780) | -0.92 (0.873) | -0.80 (0.932) | -0.09 (0.770)

2. Secondary Outcome: Number of Participants Achieving a HbA1c Value of <7% at Week 12
Time Frame: 12 weeks
Population: ITT
Measure: Number; unit: participants
Arm/Group | 75 mg LX4211 qd | 200 mg LX4211 qd | 400 mg LX4211 qd | 200 mg LX4211 Bid | Placebo qd
Number analyzed (Participants) | 56 | 58 | 57 | 57 | 57
participants | 16 | 15 | 22 | 17 | 14

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) to Week 12
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 75 mg LX4211 qd | 200 mg LX4211 qd | 400 mg LX4211 qd | 200 mg LX4211 Bid | Placebo qd
Number analyzed (Participants) | 56 | 60 | 59 | 58 | 60
mg/dL | -9.5 (27.35) | -17.4 (40.45) | -27.1 (38.48) | -26.9 (35.07) | 2.2 (45.35)

4. Secondary Outcome: Change From Baseline in Body Weight at Week 12
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 75 mg LX4211 qd | 200 mg LX4211 qd | 400 mg LX4211 qd | 200 mg LX4211 Bid | Placebo qd
Number analyzed (Participants) | 57 | 60 | 59 | 59 | 60
kg | -0.995 (3.1130) | -1.956 (2.5360) | -1.848 (1.9641) | -2.477 (2.5610) | -0.395 (1.9813)

5. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SPB) at Week 12
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 75 mg LX4211 qd | 200 mg LX4211 qd | 400 mg LX4211 qd | 200 mg LX4211 Bid | Placebo qd
Number analyzed (Participants) | 57 | 60 | 59 | 59 | 60
mm Hg | -0.123 (12.6921) | -3.878 (12.1935) | -5.746 (12.3675) | -4.452 (12.1401) | -0.283 (13.5945)

6. Secondary Outcome: Change From Baseline in Triglycerides at Week 12
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 75 mg LX4211 qd | 200 mg LX4211 qd | 400 mg LX4211 qd | 200 mg LX4211 Bid | Placebo qd
Number analyzed (Participants) | 56 | 58 | 57 | 57 | 58
mg/dL | -16.2 (84.17) | 6.6 (77.05) | -16.8 (121.90) | -16.9 (73.13) | -30.5 (201.92)

ADVERSE EVENTS:
Description: Safety population
Arm/Group | 75 mg LX4211 qd | 200 mg LX4211 qd | 400 mg LX4211 qd | 200 mg LX4211 Bid | Placebo qd
Serious Adverse Events (participants affected / at risk) | 0/57 | 1/60 | 2/59 | 0/60 | 1/60
Other Adverse Events (participants affected / at risk) | 31/57 | 34/60 | 26/59 | 26/60 | 27/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 75 mg LX4211 qd (N=57) | 200 mg LX4211 qd (N=60) | 400 mg LX4211 qd (N=59) | 200 mg LX4211 Bid (N=60) | Placebo qd (N=60)
bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 75 mg LX4211 qd (N=57) | 200 mg LX4211 qd (N=60) | 400 mg LX4211 qd (N=59) | 200 mg LX4211 Bid (N=60) | Placebo qd (N=60)
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 5 | 4 | 4
Nausea (Gastrointestinal disorders) | 5 | 3 | 6 | 2 | 3
Headache (Nervous system disorders) | 6 | 6 | 3 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 5 | 1 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1 | 3 | 3
Nasopharyngitis (Infections and infestations) | 4 | 2 | 2 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1 | 4
Sinusitis (Infections and infestations) | 3 | 3 | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 1 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 2
Pollakiuria (Renal and urinary disorders) | 3 | 1 | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institutions cannot publish any data generated from the clinical trial until Sponsor publishes such data or until 18 months have elapsed since completion of the clinical trial. Proposed publication must be provided to Sponsor at least 60 days prior to submission for publication and Sponsor has 30 days from receipt to review. Sponsor can delete any info to which it objects, Confidential Information, proprietary information or patentable subject matter from the final version of the publication.